CLINICAL TRIAL: NCT01653093
Title: Imaging of the Prostate Gland Using High Field Strength 3T MRI
Brief Title: 3-Tesla MRI in Finding Tumors in Patients With Known or Suspected Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-07042; NCI-2012-00931 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT01705028 (obsolete NCT alias)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Diagnostic (3T MRI) (Experimental): Patients undergo 3T MRI, including DCE-MRI, diffusion-weighted MRI, amide-proton-transfer MRI, and MR spectroscopy scans. Patients may undergo an additional 3T MRI scan at least 24 hours after the initial scan.
  Interventions: Procedure: 3-Tesla magnetic resonance imaging (3T MRI); Procedure: diffusion-weighted magnetic resonance imaging; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Procedure: magnetic resonance spectroscopic imaging

INTERVENTIONS:
Procedure: 3-Tesla magnetic resonance imaging (3T MRI) — Undergo 3T MRI
  Other Names: 3-Tesla MRI; 3T MRI
Procedure: diffusion-weighted magnetic resonance imaging — Undergo diffusion-weighted MRI
  Other Names: diffusion-weighted MRI
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Undergo DCE-MRI
  Other Names: DCE-MRI
Procedure: magnetic resonance spectroscopic imaging — Undergo MR spectroscopy
  Other Names: 1H-nuclear magnetic resonance spectroscopic imaging; Proton Magnetic Resonance Spectroscopic Imaging

SUMMARY:
In standard clinical care, the prostate is imaged by magnetic resonance imaging (MRI) which is a procedure to take pictures of body structures by using a strong magnetic field and radio waves. The strength of the magnet used is expressed in the unit Tesla (T); a higher Tesla number means the magnet has stronger pull. Standard magnetic resonance imaging of the prostate uses a magnet 1.5 Tesla strong as well as a specialized endorectal coil (antenna) inserted into the body due to the limitations using an external body coil at this magnet strength. MRI using a 3 Tesla magnet has a theoretical advantage over imaging at 1.5 Tesla of creating a signal twice as strong that can be received by the antennas, resulting in better pictures. The goal of this study is to make the MRI procedure more comfortable for patients by using an external coil instead of an endorectal coil. With this study, researchers also want to help patients' health care teams, the surgeons in particular. Researchers will assess the impact of prostate MRI, without an endorectal coil, done at 3 Tesla and with an external body coil on helping doctors decide which approaches to disease therapy might be best for patients as well as correlate patients' study images with all other clinical imaging

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the impact of prostate MRI, without an endorectal coil, done at 3-Tesla on surgical management. This would be performed by examining the agreement of lesion location based on the MRI compared to the lesion location based on pathology and/or surgery and local extent of the disease, i.e. involvement of contiguous organs and local lymph nodes, based on the MRI compared to the local extent based on pathology and/or surgery.

II. To test the reproducibility of functional MRI (dynamic-contrast enhanced [DCE_MRI] MRI, magnetic resonance [MR] spectroscopy and diffusion-weighted MRI).

SECONDARY OBJECTIVES:

I. To assess the usefulness of MRI data in treatment planning for radiation therapy, and to test the feasibility of amide-proton-transfer MRI in prostate cancer detection.

II. To evaluate MRI changes in prostate and tumor morphology between endorectal coil versus no endorectal coil.

III. To assess the usefulness of ex-vivo prostate specimen MRI for accurate co-registration between in-vivo MRI of the prostate and pathology slides.

OUTLINE:

Patients undergo 3-tesla (3T) MRI, including DCE-MRI, diffusion-weighted MRI, amide-proton-transfer MRI, and MR spectroscopy scans. Patients may undergo an additional 3T MRI scan at least 24 hours after the initial scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected prostate disease based on clinical data will be included in the study; patients with intermediate to high grade prostate cancer (Gleason's score >= 7 and prostate-specific antigen [PSA] of > 10ng/dl) will be referred from the outpatient clinics after evaluation by the treating physicians
* Written informed consent will be signed by the patients before the MRI based on the guidelines approved by the Ohio State University Institutional Review board
* Patients must have an estimated glomerular filtration rate of >= 30 mL/min/1.73m^2 within six weeks of the MRI to be included in the study

Exclusion Criteria:

* Patients with any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc.)
* Patients with any type of ferromagnetic bioimplant that could potentially be displaced or damaged
* Patients that have vascular or aneurysm clips, or metallic staples from a surgical procedure
* Patients with permanent tattoo eye liner (may contain metallic coloring)
* Patients that may have shrapnel imbedded in their bodies, such as from war wounds, metal workers and machinists (metallic fragments in or near eyes), severe auto accident victims
* Patients that exhibit noticeable anxiety and/or claustrophobia
* Patients who cannot adhere to the experimental protocols for any reason, or have an inability to communicate with the researcher
* Patients who have cardiac or known circulatory impairment, and/or the inability to perspire (poor thermoregulatory function)
* Patients with an estimated glomerular filtration rate of < 30 mL/min/1.73m^2 within six weeks of the MRI
* Acute or chronic severe renal insufficiency (estimated glomerular filtration rate < 30 mL/min/1.73m^2)
* Acute renal dysfunction due to the hepato-renal syndrome or in the perioperative liver transplantation period

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2007-09-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic imaging quality of the prostate at 3T high field imaging without an endorectal coil | Up to 6 years
  The primary outcome in this study is the agreement in tumor staging between pathology and 3 Tesla MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knopp, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Stress, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu